

# **Trial Statistical Analysis Plan**

c03164045 -01

**BI Trial No.:** 1289.7

Title: A multi-centre, double-blind, parallel-group, randomised

controlled study to investigate efficacy, safety and tolerability of orally administered BI 409306 during a 12-week treatment period compared to donepezil and placebo in patients with cognitive

impairment due to Alzheimer's Disease.

Investigational

**Product(s):** 

BI 409306

Responsible trial statistician(s):

Telephone:

Fax:

Date of statistical

13 JUN 2017 SIGNED

analysis plan:

Version: Final


Proprietary confidential information

© 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1 T | A DT | $\mathbf{r}$ | $\mathbf{\Omega}\mathbf{E}$ | $\mathbf{CON}$ | | TTC |
|---|---|---|---|---|---|---|
| | 4 D L | ır. | Ur ' | しいい | ITEN | 113 |

| T | ITLE P | AGE | 1 |
|---|---|---|---|
| 1 | | ABLE OF CONTENTS | |
| L | | TABLES | |
| 2 | | IST OF ABBREVIATIONS | |
| 3 | | NTRODUCTION | |
| 4 | | HANGE IN THE PLANNED ANALYSIS OF THE STUDY | |
| <b>5</b> | | | |
| 3 | 5.1 | NDPOINT PRIMARY ENDPOINT | IV |
| | 5.1 | SECONDARY ENDPOINTS | |
| | 5.2.1 | Key secondary endpoint. | |
| | 5.2.2 | • • • | |
| | 01212 | Other Secondary Chaponies Williams | 10 |
| | | | 11 |
| 6 | G | ENERAL ANALYSIS DEFINITIONS | <u>12</u> |
| | 6.1 | TREATMENTS | |
| | <b>6.2</b> | IMPORTANT PROTOCOL VIOLATIONS | 14 |
| | 6.3 | PATIENT SETS ANALYSED | |
| | 6.5 | POOLING OF CENTRES | |
| | 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| | 6.6.1 | Missing efficacy data | |
| | 6.6.2 | Missing safety data and other data | |
| | 6.6.3<br>6.6.4 | Missing AE dates and times | |
| | 6.7 | Missing plasma concentrations and pharmacokinetic parameters BASELINE, TIME WINDOWS, AND CALCULATED VISITS | |
| 7 | | LANNED ANALYSIS | |
| / | 7.1 | DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS | |
| | 7.1<br>7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| | 7.3 | TREATMENT COMPLIANCE | |
| | 7.4 | PRIMARY ENDPOINT(S) | |
| | 7.4.1 | Primary efficacy analysis | |
| | 7.4.2 | Sensitivity analyses - primary and MMRM endpoints | |
| | 7.5 | SECONDARY ENDPOINTS | |
| | 7.5.1 | Key secondary endpoint | |
| | 7.5.2 | Secondary endpoints | |
| | 7.5.3 | Sensitivity analyses - secondary endpoints | |
| | | | 24 |
| | 7.7 | EXTENT OF EXPOSURE | 25 |
| | <b>7.8</b> | SAFETY ANALYSIS | |
| | 7.8.1 | Adverse events | |
| | 7.8 | 3.1.1 Assignment of AEs to treatment | |

# **Boehringer Ingelheim**

# TSAP for BI Trial No.: 1289.7


| Proprieta | ary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more | of its affiliated companies |
|---|---|---|
| | 7.8.1.2 Analysis of other significant AEs | 25 |
| | 7.8.1.3 AE summaries | |
| | 7.8.1.4 AE summaries for disclosure | 20 |
| , | 7.8.2 Laboratory data | 20 |
| , | 7.8.3 Vital signs | |
| , | 7.8.4 ECG | 27 |
| , | 7.8.5 Others | 27 |
| | 7.8.5.1 C-SSRS | 27 |
| 8 | REFERENCES | 28 |
| 9 | ADDITIONAL SECTIONS | 29 |
| 9.1 | | |
| 9.2 | C-SSRS FDA CATEGORIES | <b>3</b> 1 |
| 9.3 | SAS CODE | 32 |
| <b>10</b> | HISTORY TABLE | 33 |

# **Boehringer Ingelheim**

TSAP for BI Trial No.: 1289.7


Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Treatment descriptions | 12 |
|---|---|---|
| Table 6.1: 2 | Definition of analyzing treatment period | 13 |
| Table 6.2: 1 | important protocol violations | 15 |
| Table 6.3: 1 | Patient sets analyzed | 19 |
| Table 6.7: 1 | Time windows for all pre/on-treatment safety visits | 21 |
| Table 6.7: 2 treatment | Time windows for on-treatment efficacy measurement scheduled for each visit | |
| Table 9.1: 1 | NTB description and scoring. | 29 |
| Table 9.2.1 | CSSRS and FDA categories | 31 |
| Table 9.3.1 | SAS Code for main analyses | 32 |
| Table 10: 1 | History table | 33 |

HPC

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2 LIST OF ARREVIATIONS

| 2 LIST OF A | BBREVIATIONS |
|---|---|
| Term D | efinition / description |
| ABCB1 | ATP-binding cassette sub-family B member 1 (gene encoding for P-gp) |
| ADCS-ADL | Alzheimer's Disease Cooperative Study/Activities of Daily |
| ADCS-MCI-ADL | ADCS-ADL for mild cognitive impairment |
| AChE-Is | Acetylcholine Esterase Inhibitors |
| AD | Alzheimer's Disease |
| ADAS-cog | Alzheimer's Disease Assessment Scale-cognitive subscale |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| APOE | Apolipoprotein E |
| AUC | Area under the Curve |
| BCRP | Breast cancer resistance protein |
| BDNF | Brain-derived neurotrophic factor |
| b.i.d | bis in die (twice a day) |
| BPM | Beats per Minute |
| CDR-SB | Clinical Dementia Rating Scale–Sum of Boxes |
| BRPM | Blinded report planning meeting |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CT | Concomitant therapy |
| CCT | Cranial Computer Tomography |
| CSF | Cerebrospinal fluid |
| Cmax,ss | Maximum measured concentration in plasma (at steady state) |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTC | Common Terminology Criteria |
| CTMF | Clinical Trial Master File |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CYP | Cytochrome |
| DAT | Dementia of Alzheimer Type |
| DMC | Data Monitoring Committee |
| DMG | Dictionary Maintenance Group |
| DNA | Deoxyribonucleic Acid |
| DM&SM | Boehringer Ingelheim Data Management and Statistics Manual |
| DRA | Drug Regulatory Affairs |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| EM | Extensive metabolizer |
| EMEA | European Agency for the Evaluation of Medicinal Products |
| EudraCT | European Clinical Trials Database |
| FAS | Full Analysis Set |
| FTA | Fluorescent treponemal antibody absorbent test |
| GCP | Good Clinical Practice |

Human Pharmacology Centre

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

HR Heart Rate

IB Investigator's Brochure ICF Informed consent form

ICH International Conference on Harmonisation

IEC Independent Ethics Committee
IM Intermediate metabolizer
IPV Important protocol violation
IRB Institutional Review Board
ISF Investigator Site File

IRT Interactive Response Technology
MCPMod Multiple Comparisons & Modelling

MedDRA Medical Dictionary for Drug Regulatory Activities

MI Multiple Imputation

MNDA Myeloid cell nuclear differentiation antigen

MMRM Mixed model repeated measures
MMSE Mini-Mental-State-Examination
MQRM Medical Quality Review Meeting
MRI Magnetic Resonance Imaging

MST Medical Subteam

NMDA-R N-methyl-D-aspartate receptor NTB Neuropsychological Test Battery

P-gp P-glycoprotein Oracle Clinical O\*C OC Observed cases Original result OR Pharmacodynamics PD Pharmacogenomic(s) PG(x)Poor metabolizer PM **POC Proof of Concept** PPS Per protocol set **PSTAT** Project Statistician Pharmacokinetic PK PM Poor metabolizers PVProtocol violation Q1 Lower quartile Q3 Upper quartile **RDC** Remote Data Capture

RDC
REP
Residual Effect Period
RPR
Rapid Plasma Reagin
q.d.
quaque die (once a day)
SAE
Serious Adverse Event
SD
Standard Deviation
SE
Standard Error

SMQ Standardised MedDRA query

SOC System organ class

## **Boehringer Ingelheim**

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

SPC Summary of Product Characteristics

TCM Trial Clinical Monitor

TDMAP Trial Data Management and Analysis PlanTime to maximum plasma

 $t_{max,ss}$  concentration (at steady state)

TESS Treatment emergent signs and symptoms

TMM Team Member Medicine
TMW Trial Medical Writer
TOC Table of contents

TS Treated Set

TSAP Trial Statistical Analysis Plan

UM Ultrarapid metabolizer

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3 INTRODUCTION

As per ICH E9, the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

SAS Version 9.4 will be used for all analyses.

## 4 CHANGE IN THE PLANNED ANALYSIS OF THE STUDY

The following changes were made:

The residual effect period (washout) is defined as 7 days, this is not mentioned in Section 7.3.3 of the CTP, but is mentioned in section 5.2.2.2 of the CTP.

The data for patients entered prior to Amendment 2 will be handled as follows:

- Donepezil data will be summarized descriptively
- All treatment naïve patients will be assigned to the "No" stratum for concurrent use of AcHEI (Yes, No).
- The data for assessments removed from the study completely, or for a specific visit due to the amendment will be summarized descriptively.

## 5 ENDPOINT

#### 5.1 PRIMARY ENDPOINT

The primary endpoint is:

The Neuropsychological Test Battery (NTB) response, defined as change from baseline in total z-score after 12 weeks of treatment.

For each patient's raw scores on each of the 9 NTB tests will be converted to the standardized z-score using the baseline means and standard deviations (SDs) for each test. The baseline means and SDs will be calculated using all randomized patients. The resultant z-scores will be averaged to obtain a total z-score, incorporating all 9 NTB tests. Change from baseline will be calculated as the post-baseline composite z-score minus the pre-treatment z-score, such that a positive change indicates an improvement from baseline. The measurements taken at Visit 3 will be considered as baseline values. Further information can be found in section 9.1.

#### 5.2 SECONDARY ENDPOINTS

#### 5.2.1 Key secondary endpoint

This section is not applicable as no key secondary endpoint has been specified in the protocol.

#### **5.2.2** Other Secondary endpoints

Secondary efficacy endpoints are the same as detailed in Section 5.1.1 of the protocol. Namely, they are the following:

Change from baseline in the ADCS-ADL (Alzheimer's Disease Cooperative Study/Activities of Daily Living) score after 12 weeks of treatment.

Change from baseline CDR-SB (Clinical Dementia Rating – Sum of Boxes) after 12 weeks of treatment

Change from baseline in ADAS-Cog11 (Alzheimer's Disease Assessment Scale cognitive subscale) total score after 12 weeks of treatment.



TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6 GENERAL ANALYSIS DEFINITIONS

## **6.1 TREATMENTS**

For regimen details refer to Section 3.1 of the CTP.

The treatments and treatment periods are defined as follows:

Table 6.1: 1 Treatment descriptions

| TPATT | Long Name | Short Name |
|-------|-----------------------|-------------|
| A | BI 409306 10 mg QD | BI 10mg QD |
| В | BI 409306 25 mg QD | BI 25mg QD |
| С | BI 409306 50 mg QD | BI 50mg QD |
| D | BI 409306 25 mg BID | BI 25mg BID |
| Е | Placebo | Placebo |
| F | Donepezil 5mg/10mg QD | Donepezil |

Table 6.1: 2 Definition of analyzing treatment period

| Label | Interval | Start Date | Start time |
|---|---|---|---|
| Screening | Screening | Date of informed consent | 00:00 |
| Placebo Run-in (PBORI) | Run-in | Date of first administration of run-in medication | Time of first<br>administration of<br>run-in medication<br>12:00 if missing |
| BI 409306 10mg QD<br>BI 409306 25mg QD<br>BI 409306 50mg QD<br>BI 409306 25mg BID<br>Placebo<br>Donepezil 5mg/10mg QD | Treatment | Date of first administration of study drug | Time of first<br>administration of<br>study drug<br>12:00 if missing |
| Post-treatment | Post-treatment | Date of last intake of study<br>drug + X+1 (see definition of<br>X below) | 00:00 |
| Post-study | Post-study | Start date = Last contact date, defined as the maximum of (Trial completion date, last study drug intake + X) +1 | 00:00 |

For safety analyses, data up to 7 days after last treatment intake will be considered as on treatment for AEs and for laboratory values. To clarify;

- Screening: starts from the date of informed consent to the date of first administration of run-in medication.
- Placebo run in period: starts from the date of first administration of run-in medication to the date of first administration of randomised study drug.
- On treatment: From the first intake of randomised study drug to last intake of randomised study drug + X days, where X=7 days for safety laboratory and AE.
- Post-treatment: From end of on-treatment period until last contact. Last contact date is defined in Table 6.1: 1. Post treatment period is not applicable for patients with last contact equal to 'last intake + X + 1 days' where X is 7 days as previously specified.
- Post study: From day after last contact defined in <u>Table 6.1: 1</u>. If period starts at end of on-treatment period then post-treatment period is not applicable.

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **6.2 IMPORTANT PROTOCOL VIOLATIONS**

Important protocol violations (IPV) affecting subjects' rights will be identified separately from those affecting analysis sets in the study report. Patients with important PVs that could potentially impact efficacy endpoints will be excluded from the PPS (Refer to Section 6.3).

The protocol violations are listed in the <u>Table 6.2: 1</u> below. They will be reviewed at Medical Quality Review Meetings (MQRMs) conducted periodically based on data accumulated during the trial. A list of protocol deviations will be discussed at the blinded report planning meeting (BRPM).

If the data show other important PVs, this table will be supplemented accordingly at MQRMs or BRPMs or through team review of the manual PV log. The decision whether a patient will be excluded from the analysis will be made at the final BRPM prior to DBL.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 important protocol violations

| Category/<br>Code | Description | Example/Comment | Excluded from PPS | Automatic<br>/Manual |
|---|---|---|---|---|
| A | Entrance criteria not met | | | |
| A1 | Inclusion criteria not met | | | |
| A1.1 | Patient younger than 55 years of age | Inclusion criteria 7 not met as specified in the protocol. | Yes | Automatic |
| A1.2 | Diagnosis of mild Alzheimer's<br>Dementia not met | Inclusion criteria 1 not met as specified in the protocol. | Yes | Automatic |
| A1.3 | Inadequate MMSE or ADAS-cog11 or CDR score | Inclusion criteria 2 not met as specified in the protocol. | Yes | Automatic |
| A1.4 | Previous or current use of AD medication requirement not met. | Inclusion criteria 6 not met as specified in the protocol. | Yes | Automatic |
| A1.5 | Inadequate education and language | Inclusion criteria 5 not met as specified in the protocol. | Yes | Automatic |
| A1.6 | Inadequate study partner reliability | Inclusion criteria 4 not met as specified in the protocol. | Yes | Automatic |
| A2 | Exclusion criteria met | | | |
| A2.1 | Alzheimer's Dementia secondary disorder | Exclusion criteria 1 met as specified in the protocol. | Yes | Automatic |
| A2.2 | Substantial concomitant cerebrovascular disease | Exclusion criteria 2 met as specified in the protocol. | Yes | Automatic |
| A2.3 | Symptomatic and unstable/uncontrolled conditions | Exclusion criteria 4 met as specified in the protocol. | Yes | Automatic |
| A2.4 | Neurological disease or other psychiatric disorder | Exclusion criteria 6 met as specified in the protocol. | Yes | Automatic |
| A2.5 | Any suicidal behavior in the past 2 years | Exclusion criteria 7 met as specified in the protocol. | No | Automatic |
| A2.6 | Any suicidal ideation of type 4 or 5 in the C-SSRS in the past 3 months | Exclusion criteria 8 met as specified in the protocol. | No | Automatic |
| A2.7 | Participation in AD study less<br>than 3 months from screening,<br>treatment for disease<br>modification or non-<br>prescription medications | Exclusion criteria 9 met as specified in the protocol. | Yes | Automatic |
| A2.8 | Known history of HIV infection | Exclusion criteria 11 met as specified in the protocol. | Yes | Automatic |
| A2.9 | Prohibited drugs within 3 months prior to study participation | Exclusion criteria 17 met as specified in the protocol. | Yes | Automatic |

Proprietary confidential information @ 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 (continued) important protocol violations

| | ategory | Description | Example/Comment | Excluded from PPS | Automatic<br>/Manual |
|---|---|---|---|---|---|
| | A2.10 | Uncompensated hearing loss | Exclusion criteria 21 met as specified in the protocol. | Yes | Automatic |
| В | | Info | rmed consent not available/not done | | |
| | B1 | Informed consent not available/not done | Informed consent date missing; no signature on ICF | Exclude from All | Automatic<br>/Manual |
| | B2 | Informed consent too late | Check if informed consent date (actual consent date) was prior or on Visit 1. Applicable to all informed consents. Date of informed consent was after the date of any study-related procedure. If patient signed the wrong version of ICF and then signed the correct version of ICF with the date after screening, it is still deemed as IPV | No | Automatic /Manual |
| C | | Tr | ial medication and randomization | | |
| | C1 | Incorrect trial medication taken | | | |
| | C1.1 | Incorrect trial medication taken during study | Any deviation. Check whether the medication packages dispensed (med. Numbers entered into RDC) has the correct content (to be seen from the med. number list that was the basis for packaging). If content was correct, the deviation will only be noted. Otherwise, the cases will be described individually and possibly excluded. In addition, check whether the dispensed packages match the randomized treatment of the patient (IRT assignment). If not, and if treated consistently throughout the trial, analyze as treated. | Yes | Automatic |
| | C2 | Randomization order not followed | | | |

Proprietary confidential information @ 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 (continued) important protocol violations

| | ategory<br>Code | Description | Example/Comment | Excluded from PPS | Automatic<br>/Manual |
|---|---|---|---|---|---|
| | implemented the randomization scheme | | E.g., the same randomization number was given to different patients or the assignment of duplicate medication numbers or incorrect medication numbers. | Yes | Manual |
| | | | Verify by comparing the medication numbers and randomization numbers from IRT. | | |
| | | | If a patient actually receives the correct medication despite the wrong kit, they will not be excluded from the PPS. | | |
| | | | Vendor to check before unblinding. | | |
| | С3 | Non-compliance with study medication | | | |
| | C3.1 | Non-compliance with study medication | Compliance < 80% or >120 % | Yes if <80% | Automatic<br>/Manual |
| D | | Concomitant medication | | | |
| | D1 | Prohibited medication use before the treatment period of the trial | To be determined on a case by case basis. | Yes | Automatic<br>/Manual |
| | D2 | Prohibited medication use during the conduct of the trial | To be determined on a case by case basis. | Yes | Automatic<br>/Manual |
| E | | ] | Trial specific protocol violations | | |
| | E1 | Negative pregnancy test result not obtained during the study participation | | No | Automatic |
| | E2 | Treatment not discontinued due to HR elevation as described in CTP section 3.3.4. | | No | Automatic |
| | E3 | Study partner change during study. | | Yes | Automatic |
| | E4 | Assessments administered by unqualified rater | | Yes | Manual |
| | E5 | C-SSRS not administered at every visit | | No | Automatic |

Table 6.2: 1 (continued) important protocol violations

| | ategory<br>ode | Description | Example/Comment | Excluded from PPS | Automatic<br>/Manual |
|---|---|---|---|---|---|
| F | | Incorr | ect timing of endpoint measurements | | |
| | F1 | Incorrect timing - assessments | | | |
| | F1.1 | Assessment order not followed | NTB not administered in order specified in CTP | Yes | Automatic |
| | F1.2 | Rater switch on primary endpoint | NTB not administered by same rater | Yes | Manual |
| | F2 | Incorrect timing – times of measurements | | | |
| | F2.1 | Assessment of NTB outside of window between visits | NTB assessment time >2 hour from Visit 3 NTB assessment time. | Yes | Automatic |

**KEY:** PPS – Per Protocol Set

#### 6.3 PATIENT SETS ANALYSED

SCR - Screened set: All patients screened for the trial, with informed consent given and who completed at least one screening procedure at Visit 1.

RS- Randomized set: This patient set includes all patients who signed the informed consent form and were also randomized, regardless whether the patient was treated with trial medication or not.

TS-Treated set: All patients who were randomized and treated with at least one dose of study drug.

FAS- Full analysis set: The full analysis set (FAS) will consist of all randomized patients who were treated with at least one dose of study drug and had a baseline and at least one post baseline on treatment primary endpoint NTB assessment (or secondary endpoint assessment). The FAS will be used for the primary analyses (and secondary analyses).

PPS- Per protocol set: All patients in the FAS without important protocol deviations that impact efficacy assessments. No analyses for the CTR are planned using the PPS set.

The SCR,RS and TS will be used to populate patient disposition and the TS will be used for demographics, baseline characteristics, treatment exposure, and safety analyses (including adverse events, laboratory measurements, vital signs, and ECG). Safety analyses will assign patients to the treatment group based on the treatment received.

If a patient erroneously receives the wrong dose of study drug, the patient's efficacy data will be analyzed in the randomized treatment group and the patient's safety data will be analyzed in the actual treatment group.

The efficacy analyses will follow the intention-to-treat (ITT) principle in assigning patients to treatment groups. I.e., efficacy analyses will be analyzed as randomized using the FAS.

If a patient receives a different study drug than randomized, this will be noted as an IPV.

Table 6.3: 1 Patient sets analyzed

| Patient set | | | | |
|--------------------|--------|--------|--------|-----|
| Class of endpoint | SCR | RS | TS | FAS |
| Primary | | | | OC |
| Secondary | | | | OC |
| Further | | | | OC |
| Safety endpoints | | | OR | |
| Disposition | $OR^1$ | $OR^1$ | $OR^1$ | |
| Demographic | | $OR^2$ | OR | |
| Baseline endpoints | | OC | | |
| Disclosure tables | OR | | OR | |

- 1) Disposition table requires multiple patient sets to populate
- 2) Additional table for clinical trial disclosure requirements

Note: For definitions of OC (Observed Case) or OR (Original Results)) refer to section 6.6.

Note that the number of patients with available data for an endpoint may differ. For details, see section 6.6.



#### 6.5 POOLING OF CENTRES

This section is not applicable because centre/country is not included in the statistical model.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Original result (OR) analysis

Original result analysis implies the analysis of data exactly as observed. OR analysis will be performed on endpoints that are not meaningful to apply any imputation rule on them for replacing the missing values.

### 6.6.1 Missing efficacy data

NTB

Details on scoring with missing items are described in <u>section 9.1</u>.

ADAS-Cog11

## TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

If a patient has 3 or fewer missing ADAS-Cog/11 items, the following algorithm will be used to compute the ADAS-Cog/11 total score:

Total score = [(total score from completed items) / (maximum total score for completed items)]\*(maximum total score[=70] for all items in the scale)

If there are more than 3 missing ADAS-Cog/11 items, ADAS-Cog/11 score will be considered missing at that time point.

#### **ADCS-ADL**

For ADCS-ADL, if <30% of the items are missing, the total score will be imputed. The sum of the nonmissing items will be prorated to the sum of total items. The imputed number will be rounded up to the nearest integer. If the nearest integer is greater than the maximum possible score, the imputed score will be equal to the maximum score. If >30% of the items are missing, the total score at that visit will be considered missing. For e.g Total score = [(total score from completed items) / (maximum total score for completed items)]\*(maximum total score = 78] for all items in the scale) Supplementary material for [8].

#### CDR-SB

If only 1 box (of 6) of the CDR is missing, the sum of the boxes will be imputed by prorating the sum from the other 5 boxes. If the score from more than 1 box is not available, the CDR-SB at that visit will be considered missing. For e.g Total score = [(total score from completed items) / (maximum total score for completed items)]\*(maximum total score[=18] for all items in the scale) Supplementary material for [16].

#### Observed cases (OC) analysis

For all efficacy endpoints using MMRM analyses, it is planned to analyze only the available data that were observed while patients were on treatment, i.e., excluding the missing data. In other words, OC analysis will be performed and missing data in this analysis will not be replaced.

The following imputation methods will be used if the rate of missing data is greater than 5%.

The method below will be used for the endpoints using ANCOVA analyses.

## Last observation carried forward (LOCF) analysis

The last observation on-treatment need not necessarily be a value selected as a visit value if multiple measurements were performed within a time window for a visit. In this case the last on-treatment value within the time window will be carried forward, while the visit value can be the value that was observed closest to the planned visit date or the first value observed in

the time window. See Table 6.7: 2 for further details.

## Baseline Observation Carried Forward (BOCF)

As part of the LOCF technique, baseline values will be carried forward if no post-baseline value is available.

#### 6.6.2 Missing safety data and other data

In general, missing data will not be imputed and only observed values will be analyzed. Data of patients who withdrew after the screening examination or were not treated will be only listed.

## 6.6.3 Missing AE dates and times

Missing or incomplete AE dates are imputed according to BI standards (see "Handling of missing and incomplete AE dates") (2).

### 6.6.4 Missing plasma concentrations and pharmacokinetic parameters

Missing data and outliers of PK data are handled according to (1).

#### 6.7 BASELINE, TIME WINDOWS, AND CALCULATED VISITS

For efficacy, the baseline is defined as the pre-treatment observation at Visit 3. All other baseline variables will be observed from Visit 1.

For laboratory safety measurements, the last values prior to study drug administration will be considered as baseline values.

The midpoint between two on-treatment visits defines the end of a time window, with the midpoint being included in the time window of the preceding visit.

| Table 6.7: 1 | Time windows | for all pre/on-treatm | nent safety visits |
|--------------|--------------|-----------------------|--------------------|
|--------------|--------------|-----------------------|--------------------|

| Visit number | Visit label | Planned days | Interval (actual days on treatment) |
|---|---|---|---|
| 1 | Screening | -28 | (-∞, PBORI-1] |
| 2 | Placebo Run-in period | -14 | [PBORI ,TREATMENT-1] |
| 3 | Baseline | 1 | [NA, 1] |
| 4a | Week 1 | 8 | [2, 11] |
| 4b | Week 2 | 15 | [12, 18] |
| 4c | Week 3 | 22 | [19, 25] |
| 5 | Week 4 | 29 | [26, 43] |
| 6 | Week 8 | 57 | [44, 73] |
| EOT | Week 12 | 85 | [74, 99] |
| FU | Follow-up | 113 | [100, Study drug stop date + 7 days] |

These time windows are defined based on the planned number of days after the date of first administration of study drug. Reasons to base the time windows on the actual treatment start date rather than the randomisation date are:

• If first intake of study drug shows a large delay by e.g. more than one week after the date of randomisation, a measurement taken four weeks after randomisation rather reflects the drug effect after three weeks than after four weeks and thus may underestimate the treatment effect at this visit.

• With large delays of the introduction of study drug after the randomisation, the time window for the first on-treatment visit could include times the patient was not yet on study drug.

Table 6.7: 2 Time windows for on-treatment efficacy measurement scheduled for each on treatment visit

| | | | Time | window |
|---|---|---|---|---|
| | | | (actual days on treatment) | |
| Visit Number | Visit label | Planned days | Start | End <sup>A</sup> |
| 3 | Baseline | 1 | NA | 1 <sup>B</sup> |
| 5 | Week 4 | 29 | 2 | 57 |
| ЕОТ | Week 12 | 85 | 58 | Study drug stop |
| | | | | date + 7 days |

A In case of premature discontinuation of the study drug an EOT Visit has to be performed. If such an EOT Visit falls into the time window of a previous visit, measurements will be assigned to this previous visit and the visit value will be determined as described below. In this case the time window for the visit that includes EOT Visit will end 7 days after the study drug stop date, including Day 7.

B Only values taken prior to the start of treatment with randomised study drug can be considered baseline values. Time windows will be used for assignment of measurements to scheduled visits.

Repeated and unscheduled efficacy and safety measurements will be

assigned to the nominal visits and listed in the subject data listing (SDL) according to the time windows described above.

If there are several safety laboratory values in one time window on treatment, the worst of these will be selected for the by-visit analyses.

For efficacy measurements, only one observation per time window will be selected for analysis at an on-treatment visit — the value will be selected which is closest to the protocol planned visit day. If there are two observations which have the same difference in days to the planned day or if there are two observations on the same day, the first value will be used. If an observation is available on the last day of treatment, this observation will be preferably selected over any later observation that is still within the time window.

Note: for LOCF imputation, the last observed on-treatment value will be carried forward, whether or not it was selected in the previous time window. For more details on LOCF refer to section 6.6.

#### 7 PLANNED ANALYSIS

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / SD / Min / Median / Max.For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles should be preferred to mean, standard deviation, minimum and maximum.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

#### 7.1 DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report.

A summary of concomitant diseases will be provided by treatment group, System Organ Class (SOC) and Preferred Term (PT).

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report.

Overall compliance will be calculated as mentioned in CTP section 4.3

#### 7.4 PRIMARY ENDPOINT(S)

The primary analysis is at 12 weeks and will be performed on the full analysis set (FAS).

Figures and tables will be displayed for the MMRM analysis results over time.

Assignment to stratum will be base on IRT and eCRF data.

#### 7.4.1 Primary efficacy analysis

The primary analysis and hypothesis testing are described in section 7.3.1 of the CTP.



## 7.5 SECONDARY ENDPOINTS

Figures and tables will be displayed for the MMRM and ANCOVA analyses results over time.

## 7.5.1 Key secondary endpoint

This section is not applicable as no key secondary endpoint has been specified in the protocol.

## 7.5.2 Secondary endpoints

The same primary analysis model will be performed for the secondary endpoint CDR-SB.

The secondary endpoints ADAS-Cog11 and ADCS-ADL will use the following model:

## ANCOVA:

Analysis of covariance will be used for the change from baseline secondary endpoint score after 12 weeks of treatment; terms include baseline value for the secondary endpoint measure, treatment and stratification factor current AChE-I use.



TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 7.7 EXTENT OF EXPOSURE

Extent of exposure will be calculated as the difference between last intake of study drug and the first administration of the study drug plus one day. Cumulative exposure will be displayed by >=weeks displayed in the CTP flowchart.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set.

Analysis will be performed as defined in Section 7.3.3 of the CTP.

#### 7.8.1 Adverse events

### 7.8.1.1 Assignment of AEs to treatment

Unless otherwise specified, the analyses of adverse events will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and NOT on the number of AEs.

For analysis multiple AE occurrence data on the CRF will be collapsed into an AE event provided that all of the following applies:

All AE attributes are identical (LLT, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome).

The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence)

For further details on summarization of AE data, please refer to (2,3)

The analysis of adverse events will be based on the concept of treatment emergent adverse events. That means that all adverse events occurring between first drug intake till last drug intake + residual effect period will be assigned to the randomized treatment. All adverse events occurring before first drug intake will be assigned to 'screening' and all adverse events occurring after the residual effect period will be assigned to 'post-treatment' (for listings only). For details on the treatment definition, see section 6.1.

#### 7.8.1.2 Analysis of other significant AEs

According to ICH E3 (11), AEs classified as 'other significant' needs to be reported and will include those non-serious and non-significant adverse events with

(i) 'action taken = discontinuation' or 'action taken = reduced', or

(ii) marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

#### 7.8.1.3 AE summaries

An overall summary of adverse events will be presented.

The frequency of patients with adverse events will be summarized by treatment, primary system organ class and preferred term (mention MedDRA levels to be displayed in the tables). Separate tables will be provided for patients with other significant adverse events according to ICH E3 (4), for patients with significant non-serious adverse events (only if these are defined for the project) and for patients with serious adverse events, for patients with AEs leading to discontinuation, and for patients with drug-related AEs.

The system organ classes will be sorted by default alphabetically, preferred terms will be sorted by frequency (within system organ class).

#### 7.8.1.4 AE summaries for disclosure

The following AE data is needed for disclosure on clinicaltrials.gov and EudraCT. This data will be included in section 16.1.9.2:

- Number of patients with non-serious AEs > of 5 %
- Total number of deaths (all causes entire study period)
- Total number of deaths resulting from drug-related adverse events
- Total number of serious adverse events
- Total number of serious adverse events related to treatment
- Total number of fatal adverse events
- Total number of fatal adverse events related to treatment

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (5).

Baseline for safety laboratory parameters will be the last available measurement before the start of randomized study drug.

Laboratory measurements taken up to 7 days after the last administration of randomised study drug will be considered as on-treatment.

Only patients with at least one available on-treatment value will be included in the analysis of an individual laboratory parameter. All individual data will be presented in listings.

Study visits will be presented by the Visit labels in Table 6.7.1,

#### 7.8.3 Vital signs

Only descriptive statistics are planned for this section of the report.

## **Boehringer Ingelheim**

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.8.4 ECG

12-lead ECG measurements will be assessed as described in the CTP Flow Chart. ECG-findings before first intake of trial drug will be considered as baseline condition. Any clinically significant new findings in the ECG measurement after the first ECG will be considered as AEs and analyzed as planned in <u>section 7.8.1</u>.

## **7.8.5** Others

#### 7.8.5.1 C-SSRS

The individual items and categories of suicidal ideation and behaviour from the C-SSRS will be summarized through descriptive statistics according to section 9.2 and [9].

## **8 REFERENCES**

- 1 001 MCS 36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON.
- 2 001-MCG-156\_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON.
- 3 001-MCG-156: "Handling and summarization of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON.
- 4 CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version
- 5 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version; IDEA for CON.
- 6 Harrison J, Minassian SL, Jenkins L, Black RS, Koller M, Grundman M, . A neuropsychological test battery for use in Alzheimer disease clinical trials. Arch Neurol 2007;64(9):1323-1329.
- Salloway S, Sperling R, Fox NC, et al. Two phase 3 trials of bapineuzumab in mild-to-moderate Alzheimer's disease. N Engl J Med 2014;370:322-33.
- 8 Doody RS, Thomas RG, Farlow M, et al. Phase 3 trials of solanezumab for mild-to-moderate Alzheimer's disease. N Engl J Med 2014;370:311-21.
- 9 001-MCG-117: "Implementation at BI of the FDA guidance on prospective assessment of suicidal ideation and behavior", current version; IDEA for CON

## 9 ADDITIONAL SECTIONS

#### 9.1 CALCULATION OF NTB TOTAL SCORE

Below is a description for the NTB along with detail on deriving the scores for the total scores and several subscales. The derivations are based on [6] and the supplementary information from [7].

## Table 9.1: 1 NTB description and scoring

The NTB is a cognitive assessment made up of the following 9 component tests:

- 1. Wechsler Memory Scale Visual Paired Associates-Immediate (WMVis-I), range 0 to 18;
- 2. Wechsler Memory Scale Verbal Paired Associates-Immediate (WMVer-I), range 0 to 24;
- 3. Rey Auditory Verbal Learning Test-Immediate (RAVL-I), range 0 to 105;
- 4. Wechsler Memory Scale-Digit Span (WMDS), range 0 to 24;
- 5. Controlled Word Association Test (COWAT);
- 6. Category Fluency Test (CFT);
- 7. Wechsler Memory Scale Visual Paired Associates-Delayed (WMVis-D), range 0 to 6;
- 8. Wechsler Memory Scale Verbal Paired Associates-Delayed (WMVer-D), range 0 to 8;
- 9. Rey Auditory Verbal Learning Test-Delayed (RAVL-D), range 0 to 30.

The first 3 tests assess immediate memory (WMVis-I, WMVer-I, RAVL-I), the second 3 assess executive function (WMDS, COWAT, CFT), and the last 3 assess delayed memory (WMVis-D,

WMVer-D, RAVL-D). Higher scores indicate better cognition on all tests.

First, a total score for each component test except the RAVL-D is calculated by summing all the scores. For the RAVL-D, the total score is calculated as:

total part 7 + total part 8 correct + (15 - total part 8 incorrect).

Then, a z-score for each component test is calculated as follows. For each subject j, at assessment time point t (with t = 0 denoting baseline), let  $y_{ijt}$  denote subject j's score at time t for the ith component test (i = 1, ..., 9). Then the corresponding z-score, denoted  $z_{ijt}$ , is defined as:

$$z_{iit} = (y_{iit} - \overline{y}_{i0}) / s_{i0}$$

## **Boehringer Ingelheim**

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Where  $y_{i0}$  and  $s_{i0}$  denote the average and the standard deviation of the baseline scores on the *i*th component test across all study subjects in the FAS.

Finally, the NTB total score  $z_{jt}$  for the *j*th subject at time t is calculated by averaging the 9 component test z-scores:

$$z_{ijt} = (z_{1jt} + \dots + z_{9jt})/9$$

The NTB total z-score will be calculated only if scores for at least 6 of the 9 component tests are not missing [6].

In addition, the following subscales are defined:

- NTB Immediate Memory z-score average of the 3 immediate memory component test zscores;
- NTB Delayed Memory z-score average of the 3 delayed memory component test z-scores;
- NTB All Memory z-score average of all 6 memory component test z-scores;
- NTB Executive Function z-score average of the 3 executive function component test zscores.

•

The Immediate Memory, Delayed Memory, and Executive Function z-scores will be calculated only if at least 2 of the 3 components tests are not missing. The All Memory z-score will be calculated only if at least 4 of the 6 components tests are not missing.

The NTB total z-score (as well as NTB Immediate Memory, NTB Delayed Memory, NTB All Memory, and NTB Executive Function z-scores) will be analyzed using the same MMRM as described for the primary analyses. These analyses will be conducted for the FAS.

# 9.2 C-SSRS FDA CATEGORIES

Eleven FDA categories and equivalent C-SSRS categories as the standard for classifying suicidal ideation and behavior

Table 9.2.1 CSSRS and FDA categories

| FDA Categories | Equivalent C-SSRS categories |
|---|---|
| Suicidal ideation: | Suicidal ideation: |
| 1. Passive | 1. Wish to be dead |
| 2. Active: Nonspecific (no method, intent, or plan) | 2. Non-specific active suicidal thoughts |
| 3. Active: Method, but no intent or plan | 3. Active suicidal ideation with any methods (not plan) without |
| | intent to act |
| 4. Active: Method and intent, but no plan | 4. Active suicidal ideation with some intent to act, without specific plan |
| 5. Active: Method, intent, and plan | 5. Active suicidal ideation with specific plan and intent |
| Suicidal behavior: | |
| 6. Preparatory actions toward imminent suicidal behaviors | Suicidal behavior: 6. Preparatory acts or behaviour |
| 7. Aborted attempt | o. Treparatory deta of benavious |
| 8. Interrupted attempt | 7. Aborted attempt |
| 9. Suicide attempt | 8. Interrupted attempt |
| 10. Completed suicide | 9. Non-fatal suicide attempt |
| | 10. Completed suicide |
| 11. Self-injurious behavior, no suicidal intent | 11. Self-injurious behavior without suicidal intent |

# 9.3 SAS CODE

The below table summarises the SAS code for the main analyses

Table 9.3.1 SAS Code for main analyses

| Analysis | Code | Comments |
|---|---|---|
| Dose response | Test the following model:<br>$\mu(d_i) = \beta_0 + \beta_1 d_i + \beta_2 d_i^2$ | Dose is treated as a continuous variable. |
| | PROC GLM DATA=one; MODEL chgept = trt trt*trt; RUN; | $\mu(d_i)$ denotes the mean response of dose level i. |
| | Treat BID dose as an in between dose = $(QD + 2*QD)/2$ | |
| MMRM | PROC MIXED DATA=dat cl method=reml ORDER=formatted; CLASS trt visit patient <achel>; MODEL chgept = trt baseline visit trt*visit baseline*visit <achel> / ddfm=KR solution; REPEATED visit / type=un subject=patient r rcorr; LSMEANS trt*visit / pdiff=all cl; RUN;</achel></achel> | current AChEI use for 1289.7 |
| ANCOVA | PROC MIXED data=one METHOD=reml ORDER=formatted; CLASS trt; MODEL chgept = baseline trt <achei>;; LSMEANS trt / CL DIFF OM; RUN;</achei> | current AChEI use for 1289.7 |

# **Boehringer Ingelheim**

TSAP for BI Trial No.: 1289.7 

Proprietary confidential information @ 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10 HISTORY TABLE

Table 10: 1 History table

| Version | Date<br>(DD-Mmm-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 13-Jun-17 | | None | This is the final TSAP without any modification |